CLINICAL TRIAL: NCT00061945
Title: A Phase I/II Dose Escalation Study of Subcutaneous Campath-1H (NSC #715969, IND #10864) During Intensification Therapy in Adults With Untreated Acute Lymphoblastic Leukemia (ALL)
Brief Title: Alemtuzumab and Combination Chemotherapy in Treating Patients With Untreated Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02807; NCI-2012-02807 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR302482; CALGB 10102 (Other: Cancer and Leukemia Group B); CALGB-10102 (Other: CTEP); U10CA031946 (NIH)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Acute Undifferentiated Leukemia; B-cell Adult Acute Lymphoblastic Leukemia; B-cell Childhood Acute Lymphoblastic Leukemia; L1 Adult Acute Lymphoblastic Leukemia; L1 Childhood Acute Lymphoblastic Leukemia; L2 Adult Acute Lymphoblastic Leukemia; L2 Childhood Acute Lymphoblastic Leukemia; Philadelphia Chromosome Negative Adult Precursor Acute Lymphoblastic Leukemia; Philadelphia Chromosome Positive Adult Precursor Acute Lymphoblastic Leukemia; Philadelphia Chromosome Positive Childhood Precursor Acute Lymphoblastic Leukemia; T-cell Adult Acute Lymphoblastic Leukemia; T-cell Childhood Acute Lymphoblastic Leukemia; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Allopurinol; Cyclophosphamide; Daunorubicin; Vincristine; Dexamethasone; Asparaginase; Filgrastim; Imatinib Mesylate; Methotrexate; Cytarabine; Trimethoprim, Sulfamethoxazole Drug Combination; Mercaptopurine; Leucovorin; Alemtuzumab; Acyclovir

ARMS (1):
- Treatment (alemtuzumab and combination chemotherapy) (Experimental): See detailed description.
  Interventions: Drug: allopurinol; Drug: cyclophosphamide; Drug: daunorubicin hydrochloride; Drug: vincristine sulfate; Drug: dexamethasone; Drug: asparaginase; Biological: filgrastim; Drug: imatinib mesylate; Drug: methotrexate; Drug: cytarabine; Drug: trimethoprim-sulfamethoxazole; Drug: mercaptopurine; Drug: leucovorin calcium; Biological: alemtuzumab; Drug: acyclovir; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: allopurinol — Given PO
Drug: cyclophosphamide — Given IV
Drug: daunorubicin hydrochloride — Given IV
Drug: vincristine sulfate — Given IV
Drug: dexamethasone — Given PO and as eye drops
Drug: asparaginase — Given SC
Biological: filgrastim — Given SC
Drug: imatinib mesylate — Given PO
Drug: methotrexate — Given IT, IV, and PO
Drug: cytarabine — Given IV
Drug: trimethoprim-sulfamethoxazole — Given PO
Drug: mercaptopurine — Given PO
Drug: leucovorin calcium — Given IV and PO
Biological: alemtuzumab — Given SC
Drug: acyclovir — Given PO
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of alemtuzumab when given together with combination chemotherapy and to see how well it works in treating patients with untreated acute lymphoblastic leukemia. Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy also work in different ways to kill cancer cells or stop them from growing. Giving alemtuzumab together with combination chemotherapy may be a better way to block cancer growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and toxicity profiles of escalating doses of Campath-1H (alemtuzumab) given subcutaneously during post-remission intensification treatment of adults with acute lymphoblastic leukemia (ALL).

II. To determine the disease-free survival (DFS) and overall survival (OS) when Campath-1H is used during post-remission intensification treatment of adults with ALL.

III. To determine whether antibody treatment with Campath-1H can further reduce minimal residual disease states in adult ALL.

IV. To obtain preliminary descriptive data on serum levels of Campath-1H during course IV, module D using limited pharmacokinetic sampling during the phase I and II components of the study.

V. To obtain feasibility data on the addition of imatinib to Cancer and Leukemia Group B (CALGB) induction and postremission combination chemotherapy for patients with Philadelphia chromosome positive (Ph+) ALL.

OUTLINE: This is a dose-escalation study of alemtuzumab.

COURSE 1 (module A): Patients receive allopurinol orally (PO) 4 times daily (QID) on days 1-14, cyclophosphamide* intravenously (IV) over 15-30 minutes on day 1, daunorubicin hydrochloride IV on days 1-3, vincristine sulfate IV on days 1, 8, 15, and 22, dexamethasone PO twice daily (BID) on days 1-7 and 15-21, asparaginase subcutaneously (SC) on days 5, 8, 11, 15, 18, and 22, and filgrastim SC on days 4-11. Patients who are Ph+ also receive imatinib mesylate PO on days 15-28.

*Note: Patients who are = 60 years old do not receive cyclophosphamide.

COURSE 2 (module B): Patients receive methotrexate intrathecally (IT) on day 1, cytarabine IV over 3 hours on days 1-3, dexamethasone as eye drops QID on days 1-4, trimethoprim-sulfamethoxazole PO BID 3 times weekly on days 1-29, and cyclophosphamide, asparaginase and filgrastim as in course 1. Patients who are Ph+ also receive imatinib mesylate PO on days 1-28.

COURSE 3 (module C): Patients receive vincristine sulfate IV on days 1, 15, and 29, methotrexate IV over 3 hours and IT on days 1, 15, and 19, methotrexate PO every 6 hours on days 1-2, 15-16, and 29-30, mercaptopurine PO on days 1-35, leucovorin calcium IV on days 2, 16, and 30, leucovorin calcium PO every 6 hours on days 3-4, and trimethoprim-sulfamethoxazole PO BID 3 times weekly on days 1-43. Patients who are Ph+ also receive imatinib mesylate PO on days 1-42.

COURSE 4 (module D): Patients receive alemtuzumab SC 3 times weekly for 4 weeks and begin acyclovir PO QID for 6 months (continuing through course 8).

* Phase I Cohort 1: 10 mg
* Phase I Cohort 2: 20 mg
* Phase I Cohort 3/Phase II MTD: 30 mg

COURSE 5 (module A): Patients repeat course 1, minus allopurinol.

COURSE 6 (module B): Patients repeat course 2.

COURSE 7 (module C): Patients repeat course 3.

COURSE 8: Patients receive mercaptopurine PO, vincristine sulfate IV on day 1, dexamethasone PO on days 1-5, methotrexate PO on days 1, 8, 15, and 22, and trimethoprim-sulfamethoxazole PO BID 3 days weekly. Patients who are Ph+ also receive imatinib mesylate PO on days 1-28. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal histologic diagnosis of precursor B or precursor T lymphoblastic leukemia (World Health Organization [WHO] classification), L1 or L2 ALL or acute undifferentiated leukemia (AUL) (French-American-British Cooperative group [FAB] Classification); Burkitt-type ALL (FAB L3, surface immunoglobulin [SIg]+) are excluded
* No prior treatment for leukemia with three permissible exceptions:

  * Emergency leukapheresis II. Emergency treatment for hyperleukocytosis with hydroxyurea III. Cranial radiation therapy (RT) for central nervous system (CNS) leukostasis (one dose only)
* All patients must have a pre-treatment bone marrow or peripheral blood sample submitted for central immunophenotyping; only those patients who express CD52 >= 10% in the leukemia blast cell channel will be eligible to receive Campath-1H during module D, course IV

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2003-06; Primary Completion 2007-12 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2003 to May 2007, a total of 302 participants were recruited.
Pre-assignment Details: Two (2) participants cancelled prior to receiving any treatment and were removed from all analyses.
Groups:
- Phase I - Alemtuzumab and Combination Chemotherapy: COURSE 1-allopurinol (ALL) orally (PO) 4x daily (QID) d1-14, cyclophosphamide (CTX) intravenously (IV) d1, daunorubicin IV d1-3, vincristine (VCR) IV d1,8,15 & 22, dexamethasone (DEX) PO 2x daily (BID) d1-7 & 15-21, asparaginase (APG) subcutaneously (SC) d5,8,11,15,18 & 22, and filgrastim (FIL) SC d4-11. Ph+ pts imatinib (IMT) PO d15-28 COURSE 2-methotrexate (MTX) intrathecally (IT) d1, cytarabine IV d1-3, DEX eye drops QID d1-4, cotrimoxazole (CRT) PO BID 3x wkly d1-29 and CTX, APG & FIL as course 1. Ph+ pts IMT PO d1-28 COURSE 3-VCR IV d1,15 & 29, MTX IV & IT d1,15 & 19, MTX PO q6 hr d1-2,15-16 & 29-30, mercaptopurine (6-MP) PO d1-35, leucovorin (LCV) IV d 2,16 & 30, LCV PO q6 hr d3-4 & CRT PO BID 3x wkly d1-43. Ph+ pts IMT PO d1-42 COURSE 4-alemtuzumab 10,20 or 30 mg SC 3x wkly q4 wk, acyclovir PO QID q6 mo COURSE 5-course 1 COURSE 6-course 2 COURSE 7-course 3 COURSE 8-6-MP PO, VCR IV d1, DEX PO d1-5, MTX PO d1,8,15 & 22 and CRT PO BID 3d wkly. Ph+ pts IMT PO d1-28 q24 mo
- Phase II - Alemtuzumab and Combination Chemotherapy: COURSE 1-allopurinol (ALL) orally (PO) 4x daily (QID) d1-14, cyclophosphamide (CTX) intravenously (IV) d1, daunorubicin IV d1-3, vincristine (VCR) IV d 1,8,15 & 22, dexamethasone (DEX) PO 2x daily (BID) d 1-7 & 15-21, asparaginase (APG) subcutaneously (SC) d 5,8,11,15,18 & 22, and filgrastim (FIL) SC d 4-11. Ph+ pts imatinib (IMT) PO d 15-28 COURSE 2-methotrexate (MTX) intrathecally (IT) d1, cytarabine IV d1-3, DEX eye drops QID d 1-4, cotrimoxazole (CRT) PO BID 3x wkly d1-29 and CTX, APG & FIL as course 1. Ph+ pts IMT PO d1-28 COURSE 3-VCR IV d 1,15 & 29, MTX IV & IT d 1,15 & 19, MTX PO q6 hr d 1-2,15-16 & 29-30, mercaptopurine (6-MP) PO d1-35, leucovorin (LCV) IV d 2,16 & 30, LCV PO q6 hr d 3-4 & CRT PO BID 3x wkly d1-43. Ph+ pts IMT PO d1-42 COURSE 4-alemtuzumab 30 mg SC 3x wkly q4 wk, acyclovir PO QID q6 mo COURSE 5-course 1 COURSE 6-course 2 COURSE 7-course 3 COURSE 8-6-MP PO, VCR IV d1, DEX PO d1-5, MTX PO d 1,8,15 & 22 and CRT PO BID 3x wkly. Ph+ pts IMT PO d1-28 q24 mo
Period: Registration Through Course 3
Arm/Group | Phase I - Alemtuzumab and Combination Chemotherapy | Phase II - Alemtuzumab and Combination Chemotherapy
Started | 119 | 181
Completed | 25 | 66
Not Completed | 94 | 115
Not completed — Not Alemtuzumab Eligible | 18 | 25
Not completed — Early discontinuation during course I-IV | 76 | 90
Period: Course IV: Alemtuzumab
Arm/Group | Phase I - Alemtuzumab and Combination Chemotherapy | Phase II - Alemtuzumab and Combination Chemotherapy
Started | 25 | 66
Completed | 18 | 50
Not Completed | 7 | 16
Not completed — Declined Alemtuzumab | 1 | 1
Not completed — Early exits | 6 | 15

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Alemtuzumab and Combination Chemotherapy; Phase II - Alemtuzumab and Combination Chemotherapy: See detailed description or participant flow.
- Total: Total of all reporting groups
Arm/Group | Phase I - Alemtuzumab and Combination Chemotherapy | Phase II - Alemtuzumab and Combination Chemotherapy | Total
Number analyzed (Participants) | 119 | 181 | 300
Age, Continuous [Median (Full Range); unit: years] | 48.3 [30.5 to 59.8] | 46.5 [29 to 58.4] | 46.8 [29 to 59.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 73 | 128
  Male | 64 | 108 | 172
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 17 | 28
  White | 101 | 150 | 251
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 9 | 11
Region of Enrollment [Number; unit: participants]
  United States | 119 | 181 | 300

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Alemtuzumab (Phase I)
Description: The maximum tolerated dose is defined as the highest alemtuzumab dose at which less than 40% of patients develop the dose limiting toxicity (DLT), where DLT is defined as the inability to proceed (due to medical complications) with the protocol treatment within six weeks of receiving the last dose of alemtuzumab. Groups of six patients will be enrolled into each cohort at the time of re-registration prior to starting Course IV. After a cohort has accrued 6 patients and at least 3 have completed the 2-6 week post alemtuzumab observation period without DLT, the incoming patients will be assigned to the next cohort in the table while the DLT and other toxicities continue to be assessed for the newly closed cohort. If less than 3 out of 6 enrolled patients in a cohort have completed the 2-6 week post alemtuzumab observation period without DLT, additional patients may continue to enroll in that same cohort, i.e., accrual will not be suspended while waiting for patient follow-up data.
Time Frame: 6 weeks
Population: Only participants who started Alemtuzumab were analyzed per study design. Specifically, one patient declined Alemtuzumab and was excluded from this analysis.
Measure: Number; unit: mg
Arm/Group | Phase I - Alemtuzumab and Combination Chemotherapy
Number analyzed (Participants) | 24
mg | 30

2. Primary Outcome: Number of Participants Who Proceed to Course V Within 2-6 Weeks of the Last Dose of Alemtuzumab (Phase II)
Description: The primary endpoint is the number of participants who are able to proceed to course V within two - six weeks of completion of course IV.
Time Frame: 8 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Phase II - Alemtuzumab and Combination Chemotherapy
Number analyzed (Participants) | 65
participants | 30

3. Secondary Outcome: Minimal Residual Disease (MRD) During Treatment With Alemtuzumab (Phase II)
Description: Minimal Residual Disease measures the presence of of circulating leukemia cells in the body. Patients that report a Complete Response (CR) during treatment are further tested to determine the presence of small amounts of circulating leukemia cells. Here we report the number of patients who were MRD negative.
Time Frame: 9 years 4 months
Population: Patients who reported a Complete Response (CR) during treatment and were analyzed for the presence of circulating leukemia cells.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II - Alemtuzumab and Combination Chemotherapy
Number analyzed (Participants) | 51
Participants | 16

4. Secondary Outcome: Disease-free Survival, for Only Complete Response Patients
Description: Disease Free Survival (DFS) is defined as the time from a Complete Response (CR) until death or relapse. The date of last clinical assesment will be used as the censor date for patients with no death or relapse. The DFS will be estimated using the Kaplan-Meier method with confidence intervals presented.
Time Frame: 9 years 4 months
Population: All patients who received protocol treatment and had a complete response (CR) during treatment were included in this analysis. Phase I patients, who achieved complete response, were included with the phase II patients, who achieved complete response, for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I - Alemtuzumab and Combination Chemotherapy | Phase II - Alemtuzumab and Combination Chemotherapy
Number analyzed (Participants) | 92 | 145
months | 58.6 [24.8 to 103.8] | 19.8 [14.3 to 28.4]

5. Secondary Outcome: Overall Survival
Description: Overall Survival is defines as the time from registration to death due to any cause. It is estimated using the Kaplan-Meier method with confidence intervals presented.
Time Frame: 9 years 4 months
Population: All patients who registered, received protocol treatment, and were eligible were evaluated for this endpoint. Phase I patients were included with the phase II patients for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I - Alemtuzumab and Combination Chemotherapy | Phase II - Alemtuzumab and Combination Chemotherapy
Number analyzed (Participants) | 116 | 181
months | 33.6 [19.8 to 72.1] | 23.1 [18.4 to 32.0]

6. Post Hoc Outcome: Number of Participants Achieving Complete Remission
Description: A complete remission (CR) requires the following: an absolute neutrophil count (segs and bands) > 1500/μl, no circulating blasts, platelets > 100,000/μl; bone marrow cellularity > 20% with trilineage hematopoiesis, and < 5% marrow blast cells, none of which appear neoplastic. All previous extramedullary manifestations of disease must be absent (e.g., lymphadenopathy, splenomegaly, skin or gum infiltration, testicular masses, or CNS involvement).
Time Frame: 9 years
Population: Three participants were deemed ineligible and excluded from this analysis.
Measure: Number; unit: participants
Groups:
- Phase I - Alemtuzumab and Combination Chemotherapy; Phase II - Alemtuzumab and Combination Chemotherapy: See detailed description
Arm/Group | Phase I - Alemtuzumab and Combination Chemotherapy | Phase II - Alemtuzumab and Combination Chemotherapy
Number analyzed (Participants) | 116 | 181
participants | 92 | 145

ADVERSE EVENTS:
Arm/Group | Phase I - Alemtuzumab and Combination Chemotherapy | Phase II - Alemtuzumab and Combination Chemotherapy
Serious Adverse Events (participants affected / at risk) | 60/119 | 98/181
Other Adverse Events (participants affected / at risk) | 99/119 | 152/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Alemtuzumab and Combination Chemotherapy (N=119) | Phase II - Alemtuzumab and Combination Chemotherapy (N=181)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 32 (35) | 44 (52)
Hemoglobin decreased (Blood and lymphatic system disorders) | 59 (86) | 92 (146)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Asystole (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 5 (6)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac pain (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular failure (Cardiac disorders) | 5 (6) | 6 (8)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 4 (5)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 5 (6) | 10 (12)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular bigeminy (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Diplopia (Eye disorders) | 0 (0) | 2 (2)
Dry eye syndrome (Eye disorders) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 1 (1) | 3 (3)
Proptosis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 3 (3)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (12) | 26 (29)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 4 (4) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 9 (11)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (15) | 21 (26)
Diarrhea (Gastrointestinal disorders) | 20 (23) | 48 (59)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 11 (11)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 10 (10)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 9 (9) | 18 (19)
Endoscopy large bowel abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 5 (5)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (4)
Intestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 13 (13) | 14 (15)
Nausea (Gastrointestinal disorders) | 28 (35) | 55 (78)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 6 (7)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (21) | 40 (53)
Chest pain (General disorders) | 3 (4) | 7 (8)
Chills (General disorders) | 9 (9) | 16 (20)
Edema limbs (General disorders) | 15 (18) | 26 (35)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 33 (42) | 54 (82)
Fever (General disorders) | 6 (7) | 25 (33)
Gait abnormal (General disorders) | 0 (0) | 2 (2)
General symptom (General disorders) | 3 (3) | 0 (0)
Ill-defined disorder (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 4 (4) | 2 (2)
Irritability (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 4 (5)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (5) | 6 (6)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 7 (7)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1) | 3 (3)
Anorectal infection (Infections and infestations) | 0 (0) | 4 (4)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 6 (6)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3)
Catheter related infection (Infections and infestations) | 6 (6) | 9 (11)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1)
Encephalomyelitis infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 1 (1)
Gingival infection (Infections and infestations) | 0 (0) | 2 (2)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 1 (1) | 4 (4)
Infectious colitis (Infections and infestations) | 3 (3) | 1 (1)
Infectious meningitis (Infections and infestations) | 1 (1) | 1 (1)
Joint infection (Infections and infestations) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 3 (3) | 4 (4)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (11) | 16 (20)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 24 (27) | 52 (68)
Sinusitis (Infections and infestations) | 2 (2) | 6 (6)
Skin infection (Infections and infestations) | 4 (4) | 9 (9)
Small intestine infection (Infections and infestations) | 1 (2) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 3 (3)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1)
Urethral infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 8 (9)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Viral hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Vulval infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 11 (12) | 24 (29)
Alanine aminotransferase increased (Investigations) | 31 (39) | 61 (83)
Alkaline phosphatase increased (Investigations) | 16 (21) | 44 (48)
Amylase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 33 (39) | 61 (82)
Blood bilirubin increased (Investigations) | 48 (54) | 59 (79)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1) | 4 (6)
Coagulopathy (Investigations) | 2 (2) | 7 (7)
Creatinine increased (Investigations) | 25 (27) | 37 (50)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 25 (25) | 40 (42)
Gamma-glutamyltransferase increased (Investigations) | 5 (7) | 2 (2)
INR increased (Investigations) | 3 (3) | 15 (22)
Laboratory test abnormal (Investigations) | 3 (3) | 4 (10)
Leukocyte count decreased (Investigations) | 9 (11) | 22 (37)
Lipase increased (Investigations) | 0 (0) | 10 (11)
Lymphocyte count decreased (Investigations) | 5 (7) | 13 (16)
Neutrophil count decreased (Investigations) | 59 (81) | 90 (137)
Platelet count decreased (Investigations) | 59 (80) | 89 (141)
Weight gain (Investigations) | 1 (1) | 3 (3)
Weight loss (Investigations) | 3 (4) | 9 (9)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 16 (18) | 32 (36)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (3) | 3 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 56 (75) | 79 (122)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (2) | 9 (12)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal tubular disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 36 (41) | 40 (63)
Serum calcium decreased (Metabolism and nutrition disorders) | 37 (45) | 52 (75)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2) | 5 (6)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (5) | 7 (8)
Serum magnesium decreased (Metabolism and nutrition disorders) | 12 (13) | 28 (33)
Serum magnesium increased (Metabolism and nutrition disorders) | 3 (3) | 19 (19)
Serum phosphate decreased (Metabolism and nutrition disorders) | 15 (15) | 19 (22)
Serum potassium decreased (Metabolism and nutrition disorders) | 24 (27) | 43 (64)
Serum potassium increased (Metabolism and nutrition disorders) | 6 (6) | 9 (12)
Serum sodium decreased (Metabolism and nutrition disorders) | 23 (27) | 35 (44)
Serum sodium increased (Metabolism and nutrition disorders) | 5 (6) | 12 (15)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (10)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 19 (21)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (9)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 5 (6) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 5 (6)
Dizziness (Nervous system disorders) | 10 (11) | 12 (13)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (5)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 13 (13) | 27 (33)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 4 (4) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 3 (3) | 3 (3)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 3 (4)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 5 (6) | 8 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (16) | 26 (36)
Seizure (Nervous system disorders) | 1 (1) | 5 (5)
Sinus pain (Nervous system disorders) | 0 (0) | 3 (3)
Speech disorder (Nervous system disorders) | 4 (4) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 5 (5)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (5) | 10 (10)
Confusion (Psychiatric disorders) | 6 (6) | 10 (11)
Depression (Psychiatric disorders) | 3 (3) | 9 (10)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (7) | 10 (10)
Psychosis (Psychiatric disorders) | 1 (1) | 3 (3)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 3 (4)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 3 (7)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (2) | 3 (4)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal failure (Renal and urinary disorders) | 6 (6) | 7 (12)
Ureteric hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 3 (3)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 21 (25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 29 (40)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 16 (22)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (12)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 10 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (9)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 14 (16)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 12 (14) | 19 (21)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 4 (7)
Hypertension (Vascular disorders) | 3 (3) | 6 (7)
Hypotension (Vascular disorders) | 16 (17) | 22 (26)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 13 (13)
Vascular disorder (Vascular disorders) | 1 (1) | 1 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Alemtuzumab and Combination Chemotherapy (N=119) | Phase II - Alemtuzumab and Combination Chemotherapy (N=181)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 7 (7) | 11 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 55 (74) | 93 (141)
Hemoglobin decreased (Blood and lymphatic system disorders) | 93 (352) | 150 (650)
Lymphatic disorder (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 5 (9)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 4 (4)
Cardiac pain (Cardiac disorders) | 2 (2) | 6 (6)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 4 (4)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 3 (7)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 6 (7)
Sinus tachycardia (Cardiac disorders) | 11 (14) | 23 (25)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (4) | 2 (2)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 5 (5)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1) | 5 (11)
Eye disorder (Eye disorders) | 1 (1) | 4 (5)
Eye pain (Eye disorders) | 1 (1) | 3 (3)
Flashing vision (Eye disorders) | 1 (1) | 2 (2)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Optic nerve edema (Eye disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 3 (3) | 5 (5)
Vision blurred (Eye disorders) | 3 (3) | 13 (15)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Watering eyes (Eye disorders) | 2 (2) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 14 (18) | 45 (57)
Anal exam abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 24 (36) | 64 (87)
Diarrhea (Gastrointestinal disorders) | 47 (63) | 80 (124)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 8 (14)
Dyspepsia (Gastrointestinal disorders) | 10 (14) | 29 (37)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 10 (10)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 22 (27) | 48 (60)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 8 (8)
Esophagitis (Gastrointestinal disorders) | 6 (6) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (2) | 3 (3)
Gastric mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (4) | 7 (10)
Gastroscopy abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 3 (4) | 11 (11)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 28 (37) | 29 (35)
Nausea (Gastrointestinal disorders) | 59 (112) | 121 (287)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 4 (4)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 7 (7)
Peritoneal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 5 (5)
Rectal pain (Gastrointestinal disorders) | 3 (3) | 9 (10)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 5 (6)
Tooth disorder (Gastrointestinal disorders) | 2 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 4 (4) | 4 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 32 (54) | 78 (142)
Chest pain (General disorders) | 4 (5) | 9 (10)
Chills (General disorders) | 19 (20) | 46 (65)
Death NOS (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 17 (27) | 49 (78)
Facial pain (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 64 (154) | 116 (272)
Fever (General disorders) | 18 (19) | 51 (76)
Flu-like symptoms (General disorders) | 1 (2) | 1 (1)
Gait abnormal (General disorders) | 2 (2) | 1 (1)
General symptom (General disorders) | 1 (1) | 4 (6)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 3 (6)
Injection site reaction (General disorders) | 19 (21) | 21 (28)
Localized edema (General disorders) | 5 (5) | 10 (10)
Pain (General disorders) | 17 (19) | 20 (22)
Visceral edema (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 6 (7) | 10 (10)
Immune system disorder (Immune system disorders) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1) | 3 (3)
Anal infection (Infections and infestations) | 2 (2) | 5 (6)
Anorectal infection (Infections and infestations) | 2 (3) | 8 (11)
Bladder infection (Infections and infestations) | 3 (3) | 4 (4)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Catheter related infection (Infections and infestations) | 16 (20) | 18 (21)
Conjunctivitis infective (Infections and infestations) | 3 (3) | 2 (2)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 2 (2)
Eye infection (Infections and infestations) | 0 (0) | 2 (2)
Gingival infection (Infections and infestations) | 3 (3) | 7 (7)
Ileal infection (Infections and infestations) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 13 (15) | 16 (20)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 2 (2) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 4 (5) | 7 (8)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 4 (5) | 3 (4)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (2) | 1 (1)
Opportunistic infection (Infections and infestations) | 2 (5) | 3 (3)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 3 (3)
Paranasal sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 2 (3)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 1 (1)
Peritoneal infection (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Phlebitis infective (Infections and infestations) | 1 (3) | 1 (1)
Pneumonia (Infections and infestations) | 10 (12) | 16 (20)
Rhinitis infective (Infections and infestations) | 2 (2) | 1 (1)
Salivary gland infection (Infections and infestations) | 1 (1) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 28 (39) | 54 (64)
Sinusitis (Infections and infestations) | 10 (10) | 16 (27)
Skin infection (Infections and infestations) | 6 (8) | 20 (23)
Small intestine infection (Infections and infestations) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 2 (2) | 6 (7)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 10 (13) | 14 (17)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1)
Urethral infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (9) | 13 (17)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (2)
Viral hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 5 (5) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 5 (7)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Intraoperative hepatobiliary injury - Gallbladder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative venous injury - Vein-superior vena cava (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ADH abnormal (Investigations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 24 (38) | 39 (64)
Alanine aminotransferase increased (Investigations) | 66 (180) | 122 (328)
Alkaline phosphatase (Investigations) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 41 (68) | 93 (163)
Amylase increased (Investigations) | 4 (4) | 9 (12)
Aspartate aminotransferase increased (Investigations) | 59 (137) | 108 (266)
Blood bilirubin increased (Investigations) | 67 (131) | 101 (174)
Blood gonadotrophin abnormal (Investigations) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 2 (5)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1)
Coagulopathy (Investigations) | 7 (7) | 8 (18)
Creatinine increased (Investigations) | 21 (30) | 40 (70)
Fibrinogen decreased (Investigations) | 57 (66) | 93 (118)
Forced expiratory volume decreased (Investigations) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 6 (7) | 3 (10)
INR increased (Investigations) | 8 (10) | 25 (48)
Laboratory test abnormal (Investigations) | 8 (10) | 9 (36)
Leukocyte count decreased (Investigations) | 19 (45) | 43 (123)
Lipase increased (Investigations) | 0 (0) | 9 (10)
Lymphocyte count decreased (Investigations) | 17 (36) | 30 (65)
Neutrophil count decreased (Investigations) | 95 (312) | 147 (575)
Platelet count decreased (Investigations) | 93 (306) | 149 (594)
Serum cholesterol increased (Investigations) | 3 (3) | 2 (2)
Vital capacity decreased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 5 (7) | 5 (6)
Weight loss (Investigations) | 10 (11) | 20 (21)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 20 (27) | 54 (80)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 91 (281) | 137 (426)
Blood uric acid increased (Metabolism and nutrition disorders) | 9 (10) | 15 (25)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 9 (10)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 54 (99) | 79 (170)
Serum calcium decreased (Metabolism and nutrition disorders) | 62 (106) | 97 (204)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (10) | 7 (8)
Serum glucose decreased (Metabolism and nutrition disorders) | 8 (11) | 20 (34)
Serum magnesium decreased (Metabolism and nutrition disorders) | 17 (26) | 43 (74)
Serum magnesium increased (Metabolism and nutrition disorders) | 15 (15) | 29 (35)
Serum phosphate decreased (Metabolism and nutrition disorders) | 19 (28) | 39 (47)
Serum potassium decreased (Metabolism and nutrition disorders) | 40 (78) | 89 (184)
Serum potassium increased (Metabolism and nutrition disorders) | 8 (9) | 21 (21)
Serum sodium decreased (Metabolism and nutrition disorders) | 39 (68) | 84 (161)
Serum sodium increased (Metabolism and nutrition disorders) | 5 (6) | 8 (9)
Serum triglycerides increased (Metabolism and nutrition disorders) | 5 (5) | 4 (5)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 25 (33)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (18) | 55 (79)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 22 (27)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 12 (13)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (9) | 15 (32)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 26 (36)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 11 (16)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 26 (38)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (6) | 0 (0)
Ataxia (Nervous system disorders) | 6 (6) | 7 (10)
Cerebrospinal fluid leakage (Nervous system disorders) | 2 (3) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 19 (27) | 38 (51)
Dysgeusia (Nervous system disorders) | 8 (9) | 11 (12)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 3 (3)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 39 (66) | 88 (181)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 3 (3)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Myelitis (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 8 (8)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 8 (10)
Peripheral motor neuropathy (Nervous system disorders) | 12 (17) | 14 (22)
Peripheral sensory neuropathy (Nervous system disorders) | 52 (129) | 83 (194)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
Sinus pain (Nervous system disorders) | 0 (0) | 2 (2)
Speech disorder (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 3 (4) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 2 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 19 (24) | 21 (44)
Confusion (Psychiatric disorders) | 5 (5) | 8 (8)
Depression (Psychiatric disorders) | 20 (22) | 26 (46)
Insomnia (Psychiatric disorders) | 15 (27) | 31 (48)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 5 (5)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 3 (7)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (1) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2) | 4 (6)
Renal failure (Renal and urinary disorders) | 3 (3) | 6 (9)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 5 (5) | 13 (14)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 4 (4)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Feminization (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovulation pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 4 (4) | 4 (5)
Vaginal mucositis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 14 (24)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 55 (102)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (37) | 48 (74)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 13 (13)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (10)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 18 (21)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (12)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (49) | 33 (57)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (12)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 8 (9) | 15 (16)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 23 (26)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 29 (37) | 65 (97)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 12 (16)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Sweating (Skin and subcutaneous tissue disorders) | 9 (10) | 31 (36)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7)
Flushing (Vascular disorders) | 2 (2) | 3 (3)
Hematoma (Vascular disorders) | 1 (1) | 4 (4)
Hemorrhage (Vascular disorders) | 2 (2) | 9 (9)
Hot flashes (Vascular disorders) | 3 (7) | 2 (8)
Hypertension (Vascular disorders) | 9 (10) | 12 (15)
Hypotension (Vascular disorders) | 14 (15) | 35 (37)
Phlebitis (Vascular disorders) | 3 (3) | 4 (4)
Thrombosis (Vascular disorders) | 4 (4) | 11 (11)
Vascular disorder (Vascular disorders) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less